# **Study Protocol**

Study ID: 2019-A02748-49

Title: Attentional Impairment in People With Epilepsy

French abbreviation study: ETAPE

**Study summary:** 

Epilepsy is one of the most common chronic neurological conditions. It leads to cognitive impairment in 20-50% of patients with a structural form.

In comparison with seizures, these cognitive disorders are a major additional factor in occupational, social and family disability. They are particularly frequent (50%) in temporal epilepsies and preferably concern memory and language skills.

The cognitive consequences of epilepsy are therefore well described in the following areas: episodic memory, language, executive functions.

Concerning attentional abilities, a recent review has highlighted the lack of work in this specific field in order to properly measure the prevalence and nature of attentional disorders in epileptic patients. Indeed, attentional abilities are often mentioned in studies, but attention is a complex domain defined by four modalities: alertness, selective attention, divided attention and sustained attention. No study systematically assesses all of these modalities.

The objective of this study is to evaluate the prevalence and nature of attentional disorders in epileptic patients compared to control subjects.

- > **Primary outcome**: To evaluate the prevalence of attentional disorders in epileptic patients compared to control subjects.
- **Secondary outcome**: Assess the nature of attentional disorders in relation to executive functions and the level of anxiety-depression.
- ➤ Main endpoint : D2 task (selective attentional task)
- ➤ Other measures: attentionnal task (see below); executive task and depression and anxiety scale (total duration: around one hour and 10 minutes)

#### **Attentional tasks description**:



#### **Divided attention**

TAP 2.2 – Divided attention

Test duration: 6 minutes



#### **Sustained attention**

TAP 2.2 – Sustained attention

Test duration: 15 minutes



# **Executives task**:

Digit span

Verbal fluencies

Inhibition task: subtest incompatibility in TAP battery

Flexibility task: subtest flexibility in TAP battery

## Scales:

Neurological Disorders Depression Inventory for Epilepsy (NDDI-E)

Generalized Anxiety Disorder (GAD-7)

## **Population**: Epileptic patients versus normal control

## The inclusion criteria for patients are:

- Patients with epilepsy, according to the Fisher et al. (2005) criteria.
- Patient with written informed consent
- Affiliation to a social security insurance
- Individuals who have received full information about the organization of the research and have not objected to their participation and the use of their data.
- Person 18 years of age and older

#### The inclusion criteria for healthy subjects are:

- Individuals who have received full information about the organization of the research and have not objected to their participation and use of their data.
- Person 18 years of age and older
- Person with no neurological and/or psychiatric history

# <u>Duration of the inclusion period</u>: 5 years

<u>Duration of subject participation</u> (2 visits): There may be a delay of up to 3 months between the inclusion visit with neurological screening and the planning of the neuropsychological assessment visit after which the subject exits the study.

<u>Total research duration</u>: 5 years and 3 months.

#### References

Fisher, R. S., Boas, W. V. E., Blume, W., Elger, C., Genton, P., Lee, P., & Engel, J. (2005). Epileptic seizures and epilepsy: definitions proposed by the International League Against Epilepsy (ILAE) and the International Bureau for Epilepsy (IBE). Epilepsia, 46(4), 470-472.

Brissart H, Forthoffer N, Maillard L. Attention disorders in Epilepsy, determinants and therapeutic strategies (2019). Revue Neurologique, Mar;175(3):135-140.

Hudson, J. M., Flowers, K. A., & Walster, K. L. (2014). Attentional control in patients with temporal lobe epilepsy. Journal of neuropsychology, 8(1), 140-146.

Wisniewski, I., Wendling, A. S., & Steinhoff, B. J. (2011). Impact of side of lesion, seizure outcome and interictal epileptiform discharges on attention and memory after surgery in temporal lobe epilepsy. Epileptic Disorders, 13(1), 27-35.

Helmstaedter, C., Kemper, B., & Elger, C. E. (1996). Neuropsychological aspects of frontal lobe epilepsy. Neuropsychologia, 34(5), 399-406.